CLINICAL TRIAL: NCT01298869
Title: The Study of Immunogenicity of Quadrivalent Vaccine Against Human Papilloma Virus (HPV) Types 6, 11, 16, and 18 (HPV-6/11/16/18) in CKD Patients
Brief Title: The Study of Immunogenicity of Quadrivalent Vaccine Against Human Papilloma Virus (HPV) Types 6, 11, 16, and 18 (HPV-6/11/16/18) in Chronic Kidney Disease (CKD) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Kearkiat Praditpornsilpa, Associted Professor, Chulalongkorn University
Other Study IDs: 2011/02_Medicine
Record Dates: First submitted 2011-02-01; First posted 2011-02-18 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Kidney Disease, Stage IV (Severe); Chronic Kidney Disease, Stage V
Keywords: CKD; HPV infection; HPV vaccine; antibodies titer
MeSH Terms: conditions — Renal Insufficiency, Chronic; Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic kidney disease: Chronic kidney disease stage IV and V
  Interventions: Biological: HPV-6/11/16/18 vaccine

INTERVENTIONS:
Biological: HPV-6/11/16/18 vaccine — HPV-6/11/16/18 vaccination 3 doses at day 1, month 2, and month 6
  Other Names: Gardasil

SUMMARY:
Clinical trials have demonstrated the efficacy of HPV-6/11/16/18 vaccination (Gardasil. Merck) 3 doses at day 1, month 2, and month 6 to lower the occurrence of high-grade cervical intraepithelial neoplasia than did those in the placebo group. The immunogenicity and efficacy of the HPV vaccine has not been proven in late stage chronic kidney disease (CKD) population. The cellular and humoral immune responsiveness of CKD population are impaired by the retention of uremic toxin due to glomerular filtration rate (GFR) reduction, the vaccination efficacy can be altered and the effective dose/schedule of the vaccine may need to be adjusted, mostly increase in CKD patients.

This study aims to investigate the immunogenicity of quadrivalent HPV-6/11/16/18 vaccination (Gardasil. Merck) by current recommended dose/schedule in CKD stage IV-V patients and compare to non-CKD patients. Although a minimal peak anti-HPV response associated with protective efficacy has not been determined, the equivalent immune response in CKD and non-CKD patients if can be demonstrated by this study should be extrapolated to the CKD population. If less immune response results, the more intense dose/schedule of the vaccine should be further studied.

DETAILED DESCRIPTION:
Up to 70% of sexually active adults will become infected with human papillomavirus (HPV) during their lifetime. HPV infection can result in anogenital cancer and genital warts. These diseases are associated with substantial morbidity and mortality. Every year, 471,000 cases of cervical cancer are diagnosed worldwide. The 5-year survival for this disease is ~70%. The incidence of HPV-related anal cancer has doubled in the last 25 years. Screening programs to detect early disease are not available. Genital warts cause significant morbidity. Therefore, a prophylactic vaccine that reduces HPV infection will greatly reduce the burden of HPV disease. This study aims to demonstrate the immunogenicity of quadrivalent HPV-6/11/16/18 vaccination (Gardasil. Merck) by current recommended dose/schedule (day 1, and month 7) in CKD stage IV-V patients and to compare the immunogenicity of the vaccine in CKD stage IV-V patients and non-CKD subjects in historical cohort data.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between the ages 18 - 26 years as of visit 1 and has GFR < 30 mL/min/1.73 m2 by Modification of Diet in Renal Disease (MDRD) equation: eGFR = 175 x serum creatinine(-1.154) x Age(-0.203) x 0.742 (if female)
2. Subject is judged to be in good physical health on the basis of medical history, physical examination, and laboratory testing.
3. Subject is able to understand study procedures and agrees to participate in the study by giving written informed consent.
4. Subject is not pregnant now (as determined by a serum pregnancy test or urine pregnancy test sensitive to 25 IU -hCG) and agrees to use effective contraception through Month 7 of the study. Effective contraception will be considered: oral contraceptives, injection or implant contraception.
5. Subject has had no temperature > 37.8 C (oral) within 24 hours prior to the first injection.
6. Subject has no history of genital/anorectal warts,

Exclusion Criteria:

1. Subject is pregnant.
2. Subject has a history of known prior vaccination with an HPV vaccine.
3. Subject has a history of severe allergic reaction (e.g., swelling of the mouth and throat, difficulty breathing, hypotension or shock) that required medical intervention.
4. Subject is allergic to any vaccine component, including aluminum, yeast, or BENZONASE.
5. Subject has received any immune globulin or blood derived products within the 3 months prior to the first injection, or plans to receive any through Month 7 of the study.
6. Subject has a history of splenectomy, known immune disorders (e.g., systemic lupus erythematosus, rheumatoid arthritis), or receiving immunosuppressives (e.g., substances or treatments known to diminish the immune response such as radiation therapy, administration of antimetabolites, antilymphocytic sera, systemic corticosteroids). Individuals who have received periodic treatments with immunosuppressives, defined as at least 3 courses of oral corticosteroids each lasting at least 1 week in duration for the year prior to enrollment, will be excluded. Subjects using topical steroids (i.e., inhaled, nasal, or topical) will be eligible for vaccination.
7. Subject is immunocompromised or has been diagnosed as having HIV infection.
8. Subject has a known thrombocytopenia or other coagulation disorder that would contraindicate intramuscular injections.
9. Subject has a history of recent (within 1 year from the date of enrollment) or ongoing alcohol abuse or other drug abuse.
10. Subject is unable to give informed consent.
11. Subject has any prior history of genital/anorectal warts

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Chronic kidney disease stage IV and V population
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Titers of neutralizing antibodies for each HPV type | Day 1 (baseline) and month 7
  The geometric mean titers of neutralizing antibodies for each HPV type at day 1and month 7
Seroconversion rate | Day 1 (baseline) and month 7
  The seroconversion rate by vaccination will be calculated.

SECONDARY OUTCOMES:
Titer of neutralizing antibody of each HPV type | Day 1 (bseline) and month 7
  The neutralizing antibodies titer between CKD stage IV-V and non-CKD subjects in case-match historical cohort will be analyzed.
seroconversion rate | day 1 (baseline) and month 7
  The conversion rate by vaccination between CKD stage IV-V and non-CKD subjects in case-match historical cohort will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Kearkiat Praditpornsilpa, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn Memorial Hospital, Bangkok, Thailand